CLINICAL TRIAL: NCT00685789
Title: Study of Effects of Deqi and Neuropsychological Factors on Acupuncture Effects in Treatment of Bell's Palsy
Brief Title: Acupuncture With Deqi And Psychological Effects in Treatment of Bell's Palsy
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Hubei Hospital of Traditional Chinese Medicine (Other); Wuhan No.1 Hospital (Other); Xiangyang No.1 People's Hospital (Other); Renmin Hospital of Wuhan University (Other); Fudan University (Other); Second Affiliated Hospital of Zhengzhou University (Other); Yichang Hospital of Traditional Chinese Medicine (Other); The First Hospital of Hebei Medical University (Other); Wuhan General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Wei Wang, Department of Neurology of Tongji Hospital, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006CB504502
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2008-06

CONDITIONS: Bell's Palsy
Keywords: Bell's palsy，deqi，acupuncture, neuropsychology
MeSH Terms: conditions — Bell Palsy | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture with Deqi (Experimental): Needles were inserted and manipulated manually using the techniques such as lifting, thrusting, and twirling, until the internal compound sensation of soreness, numbness, fullness, aching, cool, warmth, heaviness and radiating sensation (Deqi) occurred. The needles were retained for 30 min.
  Interventions: Device: acupuncture, deqi
- Acupuncture without Deqi (Active Comparator): Needles were simply inserted and retained for 30 min, without any other stimulation.
  Interventions: Device: acupuncture Non-manipulation

INTERVENTIONS:
Device: acupuncture, deqi — Immediately after insertion of a needle, it is manually rotated backwards and forwards to induce the deqi sensation.
  Other Names: Manipulation
  Arms: Acupuncture with Deqi
Device: acupuncture Non-manipulation — After insertion of a needle, no manipulation is applied, and the needle is retained for 30 minutes.
  Other Names: Non-Manipulation
  Arms: Acupuncture without Deqi

SUMMARY:
The purpose of this study is to observe the influence of Deqi and neuropsychological factors on effects of acupuncture treatment for Bell's Palsy.

DETAILED DESCRIPTION:
Through long-term clinical practice，acupuncture treatment on facial paralysis has been generally proved effective；the large number of ancient and modern medical literature also have suggested that acupuncture is beneficial for facial paralysis. However,a scientific basis is still needed to be established to make sure the efficacy of acupuncture be recognized internationally.This study will adopt a series of international practice scales ,such as House Brackmann Scale,Facial Disability Index(FDI),World Health Organization Quality of Life-BREF (WHOQOL-BREF), Cattell Personality Factors (16PF),and Cancellation test to evaluate the role of deqi and neuropsychological factors in the acupuncture treatment for Bell's Palsy.

ELIGIBILITY:
Inclusion criteria:

1. Patients who were diagnosed to have unilateral facial-nerve weakness without any identifiable causes within 168 hours after onset of symptoms;
2. aged 18 to 65 years.

Exclusion criteria：

1. illiterate;
2. the facial paralysis is caused by herpes zoster;
3. recurrent facial paralysis;
4. noticeable asymmetry of the face before the illness which may affect the evaluation;
5. history of peptic ulcer disease, severe hypertension, uncontrolled diabetes, liver and kidney dysfunction, pregnancy, mental illness, or serious systemic diseases which may affect the treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
House-Brackmann scale (HBS) | 6 months after onset of symptoms

SECONDARY OUTCOMES:
facial disability index (FDI) | 6 months after onset of symptoms
World Health Organization Quality of Life-BREF(WHOQOL-BREF) | 6 months after onset of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Institute of Integrated Traditional Chinese and Western Medicine, Wuhan, Hubei, China

REFERENCES:
- [Derived] Xu SB, Huang B, Zhang CY, Du P, Yuan Q, Bi GJ, Zhang GB, Xie MJ, Luo X, Huang GY, Wang W. Effectiveness of strengthened stimulation during acupuncture for the treatment of Bell palsy: a randomized controlled trial. CMAJ. 2013 Apr 2;185(6):473-9. doi: 10.1503/cmaj.121108. Epub 2013 Feb 25. PMID 23439629